CLINICAL TRIAL: NCT06882135
Title: A Phase I Open-Label, Dose-Escalation and Dose-Expansion Trial Evaluating Safety, Pharmacokinetics, and Efficacy of HW071021 in Patients With Advanced Solid Tumors
Brief Title: HW071021 Monotherapy in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan Humanwell Innovative Drug Research and Development Center Limited Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RFSO-2024-11
Record Dates: First submitted 2025-03-07; First posted 2025-03-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HW071021 Dose Escalation (Experimental): Six dose levels were pre-specified, with a starting dose of 50 mg/day; subsequent levels may be adjusted based on pharmacokinetic (PK) and safety data.
  Interventions: Drug: HW071021 Tablets
- HW071021 Dose Expansion (Experimental): Based on the results of the dose escalation phase, 1-2 dose levels were selected.
  Interventions: Drug: HW071021 Tablets

INTERVENTIONS:
Drug: HW071021 Tablets — Administered orally at pre-specified doses once or twice daily.

SUMMARY:
This is a Phase I open-label study that will evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of HW071021 monotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This trial is an open-label, dose-escalation/expansion first-in-human study of HW071021, divided into two phases:

Phase 1 (Dose Escalation): This phase plans to enroll patients with advanced solid tumors who have no standard treatment, have failed standard treatment, or are ineligible for standard treatment. Patients will receive oral monotherapy with HW071021 at pre-specified escalating doses (single-dose and continuous-dose administration). The objectives are to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of HW071021 in patients. Selected subjects in Phase 1 will undergo a QT/QTc study to assess the drug's effects on QT/QTc intervals and cardiac safety.

Phase 2 (Dose Expansion): This phase intends to enroll patients with advanced solid tumors who have no standard treatment, have failed standard treatment, or are ineligible for standard treatment. Patients will receive continuous administration of HW071021 to provide additional clinical data for determining the Phase 2 recommended dose (P2RD) and potential indications.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older, applicable to both males and females.
2. Patients with histologically and/or cytologically confirmed recurrent and/or metastatic advanced solid tumors, mainly covering non - small cell lung cancer, colorectal cancer, pancreatic cancer, cholangiocarcinoma, and other cancer types that investigators believe may bring benefits. The selection of cancer types in the dose - expansion phase will be decided based on the data from the dose - escalation phase.
3. No standard treatment is accessible, standard treatment has failed, or the patient is not suitable for standard treatment.
4. The expected survival time is ≥ 12 weeks.
5. Participant must have adequate main organ function.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score is 0 or 1.
7. According to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, there is at least one measurable target lesion.
8. Participants who are capable of having children must agree to use two medically approved effective contraceptive methods during the study and for 6 months after the last dose. Women of childbearing age must have a negative serum pregnancy test within 7 days before dosing.
9. Have a full understanding of this study, voluntarily sign the informed consent form, and be able to follow the study's operating procedures and requirements for follow - up examinations.

Exclusion Criteria:

1. Known allergy to the investigational drug, drugs with the same mechanism of action or excipients.
2. Prior treatment with drugs targeting the same molecular target.
3. Use of other investigational drugs within 28 days before the first dose or at least 5 half - lives of the respective drug (whichever is shorter).
4. Receipt of surgery, chemotherapy, radiotherapy, targeted therapy, endocrine therapy, biological therapy, immunotherapy, anti - tumor herbal medicine, or other anti - cancer treatments within 28 days before the first dose or at least 5 half - lives of the respective drug (whichever is shorter).
5. Use of any drugs likely to interfere with trial safety within 2 weeks before dosing or at least 5 half - lives of the respective drug (whichever is shorter), and planned use during the study, including strong inhibitors/inducers of hepatic metabolic enzymes and P - gp, or substrates of hepatic metabolic enzymes with narrow therapeutic indices.
6. Undergoing major surgery within 28 days before the first dose.
7. Presence of ≥ Grade 2 toxicity from prior anti - cancer treatment (per Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0), except for toxicities deemed non - safety - critical by the investigator (e.g., alopecia, pigmentation, specific laboratory abnormalities).
8. Severe cardiovascular or cerebrovascular diseases.
9. History of clinically significant QTc interval prolongation, or QTc interval > 470 ms in females and > 450 ms in males at screening.
10. Uncontrolled/clinically symptomatic central nervous system metastases.
11. Positive for hepatitis B surface antigen (HBsAg) (except for hepatocellular carcinoma patients) with HBV DNA > 1000 IU/mL; positive for hepatitis C virus (HCV) antibody with HCV RNA positive; positive for human immunodeficiency virus (HIV) antibody; or active syphilis (positive for both TPPA and RPR).
12. Diagnosis of autoimmune disease, immunodeficiency disorder, history of organ transplantation, or planned organ transplantation.
13. Inability to swallow oral formulations and/or gastrointestinal disorders that may interfere with drug absorption.
14. Presence of any severe, uncontrolled clinical issues (e.g., uncontrolled malignant pleural effusion, ascites, pericardial effusion, or unstable psychiatric conditions) deemed unsuitable for study participation by the investigator.
15. Any significant clinical or laboratory abnormalities affecting safety assessment, as determined by the investigator.
16. Severe pulmonary diseases at screening, including pulmonary embolism, interstitial lung disease, active pulmonary infection, or other active infections deemed unsuitable for study entry by the investigator.
17. History of alcohol abuse or substance dependence.
18. Pregnant or lactating females, or females planning to become pregnant or breastfeed during the study.
19. Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetic Parameter：Maximum Plasma Concentration (Cmax）(Phase 1 only) | Up to 5 weeks
Pharmacokinetic Parameter：Area Under the Curve from Time 0 to the Last Quantifiable Data Point (AUC0-t）(Phase 1 only) | Up to 5 weeks
Pharmacokinetic Parameter：Area Under the Curve Over a Dosing Interval (AUCss,0-tau）(Phase 1 only) | Up to 2 years
Pharmacokinetic Parameter：Trough Concentration (Ctrough） | Up to 2 years
Number of patients with Dose-limiting Toxicities (DLTs) during the DLT assessment period(Phase 1 only) | Up to 5 weeks
Maximum tolerated dose (MTD) based on number of DLTs (Phase 1 only) | Up to 5 weeks
Phase II recommended dose | Up to 2 years
(C-ΔQTc) analysis (Phase 1 only) | Up to 2 years
Preliminary Efficacy：Objective Response Rate (ORR) | Up to 2 years
Preliminary Efficacy：Progression-Free Survival (PFS) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The decision not to share IPD is based on ethical and legal considerations to protect participant privacy and confidentiality. The trial involves sensitive data that, if de-identified, could still pose risks to participants in accordance with the Regulations of the People's Republic of China on the Administration of Human Genetic Resources. Additionally, the study protocol and informed consent form did not explicitly state that data would be shared beyond the trial team.